CLINICAL TRIAL: NCT07105579
Title: Effectiveness and Safety of Blinatumomab and Donor Lymphocyte Infusion in Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for High-risk Ph Negative B Cell Acute Lymphoblastic Leukemia：Phrase II, Exploratory Study
Brief Title: Effectiveness and Safety of Blinatumomab and Donor Lymphocyte Infusion in Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for High-risk Ph Negative B Cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU-HSCT-BITEDLI
Record Dates: First submitted 2025-07-15; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Leukemia; Relapse
Keywords: hematopoietic stem cell transplantation; Blinatumomab; Donor Lymphocyte Infusion; Ph negative B cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia; Recurrence | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinatumomab and Donor Lymphocyte Infusion (Experimental)
  Interventions: Drug: BITE and DLI

INTERVENTIONS:
Drug: BITE and DLI — Blinatumomab dosage:
  Cycle 1 (starting at day 60 post-transplant):Days 1-3: 9 μg/day，Days 4-14: 28 μg/day Cycles 2-4:Days 1-14: 28 μg/day Administration method: Continuous 24-hour intravenous infusion, one cycle every 3 months.
  DLI eligibility criteria:No history of grade III-IV acute GVHD (aGVHD).No active aGVHD or chronic GVHD (cGVHD) at the time of infusion
  DLI dosage:Administered at day 120 post-HSCT, CD3+ cell dose: 1 × 10⁷/kg

SUMMARY:
A single-arm trial to evaluate the effectiveness and safety of Blinatumomab and Donor Lymphocyte Infusion in maintenance therapy after allogeneic hematopoietic stem cell transplantation for high-risk Ph negative B cell acute lymphoblastic leukemia

DETAILED DESCRIPTION:
Currently, the treatment for Philadelphia chromosome (Ph)-negative adult B-cell acute lymphoblastic leukemia (B-ALL) primarily relies on traditional multi-agent combination chemotherapy. Clinical efficacy is closely associated with patient age, genetic characteristics, chemotherapy sensitivity, and minimal residual disease (MRD) status post-remission. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains the most critical curative approach for Ph-negative B-ALL. However, high-risk patients, such as those with refractory/relapsed B-ALL or MRD positivity before transplantation, exhibit significantly higher post-transplant relapse rates, reported at approximately 48%-59%, with a disease-free survival rate of less than 40%.

Multiple studies have reported that blinatumomab achieves complete remission rates of 33-50% in refractory/relapsed Ph-negative B-ALL. Previous research has shown that post-transplant blinatumomab is well-tolerated, with no treatment-related mortality, and the most common severe adverse event being cytopenia. The efficacy of blinatumomab as post-transplant prophylactic therapy depends on T-cell function.

Donor lymphocyte infusion (DLI) is widely used for the prevention and treatment of relapse after allo-HSCT. The investigators prior matched case-control study demonstrated that prophylactic DLI could reduce relapse and improve survival in high-risk acute leukemia patients after haploidentical peripheral blood stem cell transplantation. DLI products are rich in T lymphocytes, which can reverse T-cell exhaustion by altering the composition of cellular subsets in the patient's body, thereby exerting an anti-leukemic effect.

Based on the above rationale, the investigators are conducting this clinical study: a single-arm, phase II, multicenter trial to evaluate the efficacy and safety of blinatumomab combined with donor lymphocyte infusion as maintenance therapy in high-risk Ph-negative B-ALL patients after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-65 years (inclusive), regardless of gender.
2. Newly diagnosed B-ALL with CD19 expression on leukemic cells (regardless of CD19 positivity rate).
3. Ph-negative B-ALL with high-risk features post-allo-HSCT .
4. ≥2 months post-transplant with hematopoietic reconstitution.
5. Bone marrow morphology in remission and MRD-negative before enrollment.
6. ECOG performance status <3 and Karnofsky score ≥70.
7. No history of grade III/IV graft-versus-host disease (GVHD) and no active GVHD at enrollment.
8. Adequate organ function:AST and ALT ≤3× upper limit of normal (ULN), total bilirubin ≤2×ULN.Serum creatinine ≤2×ULN or creatinine clearance ≥50 mL/min (calculated by Cockcroft-Gault formula).Left ventricular ejection fraction (LVEF) ≥50% by echocardiography (ECHO).
9. Expected survival >3 months.
10. Voluntary provision of written informed consent, with ability to understand and comply with study requirements.

Exclusion Criteria:

1. History of hypersensitivity or severe adverse reactions to the study drug or structurally similar compounds, as assessed by the investigator to preclude participation.
2. Pregnant or lactating women, or women of childbearing potential unwilling to use effective contraception.
3. Severe cardiac dysfunction, including:Left ventricular ejection fraction (EF) <60%.Clinically significant arrhythmias (e.g., ventricular tachycardia, atrial fibrillation, second-degree heart block).Prolonged QTc interval (men >450 ms; women >470 ms).Myocardial infarction within the past year.Symptomatic coronary artery disease requiring medication.
4. Severe pulmonary dysfunction (obstructive and/or restrictive ventilatory impairment).
5. Severe hepatic impairment:ALT or total bilirubin (TBIL) >3× upper limit of normal (ULN).
6. Severe renal impairment:Serum creatinine (Cr) >2× ULN.24-hour creatinine clearance (Ccr) <50 mL/min.
7. Active infection or uncontrolled bleeding, as assessed by the investigator to preclude safe administration of the study drug.
8. History of thrombosis, embolism, cerebral hemorrhage, or other significant vascular events within the past year.
9. Psychiatric disorders or other conditions that impair the ability to provide informed consent or comply with study procedures.
10. Major organ surgery within the past six weeks.
11. Drug abuse or chronic alcoholism that may interfere with study assessments.
12. Prior organ transplantation (excluding hematopoietic stem cell transplantation).
13. Other conditions deemed by the investigator to make the patient unsuitable for participation.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The 2-year leukemia-free survival (LFS) after allo-HSCT. | 2 years

SECONDARY OUTCOMES:
The 2-year overall survival（OS） | 2 years
  2-year overall survival from transplant
The 2-year cumulative incidence of relapse | 2-years
The 2-year cumulative incidence of non-relapse mortality(NRM) | 2-years

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No